CLINICAL TRIAL: NCT00627731
Title: Phase 4, Randomized Study of Oral Glucocorticosteroid Administration in the Treatment of Acute Severe Asthma Exacerbation in Hospitalized Patients
Brief Title: Oral Glucocorticosteroid in the Treatment of Severe Asthma Exacerbation in Hospitalized Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hamamatsu University (Other)
Responsible Party: Principal Investigator, Naoki Inui, Department of Respiratory Medicine, Hamamatsu University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Hamamatsu-18-68; Hamamatsu-1968
Record Dates: First submitted 2008-02-22; First posted 2008-03-03 (Estimated); Last update posted 2011-09-07 (Estimated); Status verified 2009-10

CONDITIONS: Asthma
Keywords: Asthma Patients
MeSH Terms: conditions — Asthma | interventions — Methylprednisolone Hemisuccinate; Prednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): mPSL 240 mg per day for 5 days
  Interventions: Drug: methylprednisolone sodium succinate (mPSL)
- 2 (Experimental): PSL 40mg per day for 10 days
  Interventions: Drug: prednisolone (PSL)

INTERVENTIONS:
Drug: methylprednisolone sodium succinate (mPSL) — mPSL IV 240mg per day for 5 days and oral PSL 40mg per day for 5 days
  Other Names: methlyprednisolone sodium succinate
  Arms: 1
Drug: prednisolone (PSL) — PSL 40 mg per day for 10 days
  Other Names: prednisolone
  Arms: 2

SUMMARY:
A comparison of oral prednisolone administration with intravenous methylprednisolone infusion in the treatment of acute asthma exacerbation in hospitalized patients. Oral glucocorticosteroids administration may be effective as intravenous high-dose methylprednisolone infusion.

ELIGIBILITY:
Inclusion Criteria:

* Asthma patients, who need hospitalized treatment, who do not respond with initial treatment including bronchodilator and IV methylprednisolone therapy

Exclusion Criteria:

* Need for incubation
* With severe complications
* Received systemic glucocorticosteroid therapy in the previous 4 weeks

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2007-06; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Efficacy of oral prednisolone for the treatment of acute asthma | three-year

SECONDARY OUTCOMES:
The safety of oral prednisolone for the treatment of acute asthma | three-year

CONTACTS AND LOCATIONS:
Overall Officials: Kingo Chida, MD,PhD, Study Chair — Hamamatsu University
Locations (1):
- Hamamatsu University School of Medicine, Hamamatsu, Japan